CLINICAL TRIAL: NCT02179619
Title: A Randomized, Multi-center, Patient & Evaluator-blind, Matched Pairs, Active-controlled Design Clinical Study to Evaluate the Efficacy and Safety of Injection With Dermalax(Deep) as Compared to Restylane® in Correction of Nasolabial Fold
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of Dermalax(Deep) in Correction of Nasolabial Folds
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Across Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HG-HADNSF-12103
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Correction of Nasolabial Folds

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Dermalax(Deep) (Experimental): subject injected in one nasolabial fold (NLF) of one side of their face (blinded, split-face study design) in the Initial Treatment period
  Interventions: Device: Dermalax(Deep); Device: Restylane
- Restylane (Active Comparator): Subject injected in one nasolabial fold (NLF) of one side of their face (blinded, split-face study design) in the Initial Treatment period
  Interventions: Device: Dermalax(Deep); Device: Restylane

INTERVENTIONS:
Device: Dermalax(Deep) — Dermalax(Deep) injection into one nasolabial fold (NLF) of one side of the face (blinded, split-face study design) in the Initial Treatment period
Device: Restylane — Restylane Injection into one nasolabial fold (NLF) of one side of the face (blinded, split-face study design) in the Initial Treatment period

SUMMARY:
The study is to verify that Dermalax (Deep) is not inferior to the reference device, Restylane®, in terms of efficacy and safety in the correction of nasolabial folds. Subjects who voluntarily signed the informed consent and are judged to be eligible for this study will be intradermally injected both of study device and comparator device. Subjects will be randomized to receive injection of study device and comparator device on their each nasolabial fold. Efficacy is evaluated based on the change in Wrinkle Severity Rating Scale (WSRS) from baseline. Safety will be assessed based on 24 weeks follow up visits and subject diary which will be given to subjects during the first 2 weeks after the injection. Any uncomfortable things and adverse events will be investigated from subject diary and follow up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects no younger than 30 and no more than 65 years of age.
2. Subjects who scored 3 or 4 on the Wrinkle Severity Rating Scale (WSRS) and want to improve the appearance of their nasolabial folds (the subject does not need to have the same score on both sides.*)

   *The scores need not to be same on both sides, but the two nasolabial folds should have symmetry in the range of 3-4.
3. Subjects who have symmetric nasolabial folds.
4. Subjects who agreed to discontinue the use of any dermatological procedure or therapy, including facial wrinkle reduction procedures.
5. Subjects with the ability to understand and follow the instructions and who are committed to availability for the entire study period.
6. Subjects who have voluntarily decided to participate in this study and who have signed the informed consent form.

Exclusion Criteria:

1. Subjects who show hypersensitive skin reaction to the investigational devices, confirmed by the intradermal reaction test performed at screening.
2. Subjects who received an antithrombotic agent within 2 weeks prior to screening (with the exception of low dose Aspirin 100 mg, maximum of 300 mg/day) or NSAIDs or Vitamin E within 1 week.
3. Subjects with a liver problem and/or blood coagulation defect or subjects who require the administration of an antithrombotic agent during the clinical trial period (with the exception of low dose Aspirin 100 mg, maximum of 300 mg/day).
4. Subjects who have used a local ointment on their faces (medication such as steroid or retinoid are included and cosmetic products are excluded from this criterion) within 4 weeks prior to screening or subjects who are planning on using such an ointment during the clinical trial period.
5. Subjects who have received treatment for wrinkles or acne within 24 weeks prior to screening.
6. Subjects who have received facial (chemical) peels and/or skin rejuvenation procedures or plastic surgeries, including the injection of the Botulinum toxin, within 24 weeks prior to screening.
7. Subjects who have a permanent skin expander such as soft form or silicon implanted in the face.
8. Subjects who have scars on the face requiring a medical treatment but who have not received any treatment for more than a year or subjects who have scars or wounds on which the test investigational devices will be applied.
9. Subjects with skin disease or wound infection on the face.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Wrinkle Severity Rating Scale(WSRS) evaluation | at week 24
  Wrinkle Severity Rating Scale(WSRS) evaluation at week 24

SECONDARY OUTCOMES:
The mean of the WSRS scores from both the Dermalax (Deep) group and the Restylane® group | at week 8~ 48
  Wrinkle severity system scale(WSRS) evaluation at week8, week 16, week 36, week 48 by independent evaluator
The mean of the WSRS scores from both the Dermalax (Deep) group and the Restylane® group | at week 8~ 48
  Wrinkle severity system scale(WSRS) evaluation at week8, week 16, week 24, week 36, week 48 by investigator
The mean of the Global Aesthetic Improvement Scale(GAIS) scores from both the Dermalax (Deep) group and the Restylane® group | at week 8~48
  Global Aesthetic Improvement Scale(GAIS) evaluation at week8, week 16, week 36, week 48 by investigator
Mean of the Global Aesthetic Improvement Scale(GAIS) scores from both the Dermalax (Deep) group and the Restylane® group | at week 8~48
  Global Aesthetic Improvement Scale(GAIS) scores evaluation at week 8, 16, 24, 36, 48 by subjects
The proportion of subjects whose WSRS scores decreased at least 1 level | at week 0~48
  the proportion of subjects whose Wrinkle severity system scale(WSRS) scores decreased at least 1 level at week 24, 36, 48 by independent evaluator.
The proportion of subjects whose WSRS scores decreased at least 1 level | at week 0~48
  the proportion of subjects whose Wrinkle severity system scale(WSRS) scores decreased at least 1 level at week 24, 36, 48 by investigator

CONTACTS AND LOCATIONS:
Overall Officials: Beom Joon Kim, PhD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Jong Hoon Lee, PhD, Principal Investigator — Eulji General Hospital
Locations (2):
- South Korea (2):
  - Chung-ang University Hospital, Seoul
  - Eulji General Hospital, Seoul